CLINICAL TRIAL: NCT01430143
Title: Physical Activity for a Long and Healthy Life - Project FINE
Brief Title: Physical Activity for a Long and Healthy Life
Acronym: FINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Universitetssenteret på Kjeller (Other); Center for Healthy Aging (Unknown); The Novo Nordic Foundation (Other); Copenhagen University Hospital, Denmark (Other); Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Bente Merete Stallknecht, Associate professor, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: FourINonE
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Overweight; Insulin Resistance; Diabetes Mellitus, Type 2
Keywords: Exercise
MeSH Terms: conditions — Overweight; Insulin Resistance; Diabetes Mellitus, Type 2; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 600 kcal/day (Experimental): Exercise combusting 600 kcal/day, 7 days/week for 12 weeks.
  Interventions: Behavioral: Exercise
- 300 kcal/day (Experimental): Exercise combusting 300 kcal/day, 7 days/week for 12 weeks.
  Interventions: Behavioral: Exercise
- Sedentary (No Intervention): Continued sedentary living.

INTERVENTIONS:
Behavioral: Exercise — Daily exercise for 12 weeks.
  Arms: 300 kcal/day; 600 kcal/day

SUMMARY:
The aim of the study is to 1) delineate the molecular mechanisms behind the large variation in insulin sensitivity among apparently healthy subjects and to 2) establish the dose-response relationship between physical training and a) metabolic health, b) appetite and c) cultural health.

ELIGIBILITY:
Inclusion Criteria:

* Healthy according to interview
* Caucasian
* Sedentary, Vo2max < 45 ml/kg/min
* BMI 25-30 kg/m2
* Fat percentage 25% <
* Weight stable (+/- 2 kg within past 6 months)

Exclusion Criteria:

* First degree relatives with type 2 diabetes
* Hemoglobin concentration < 8 mmol/l
* Fasting plasma glucose 6.1 mmol/l <
* Blood pressure 140/90 mmHg <
* Regular intake of medicine

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in insulin sensitivity at 12 weeks | At baseline and 12 weeks
  As measured by a hyperinsulinemic, isoglycemic clamp combined with skeletal muscle and adipose tissue biopsies as well as low-dose PET/CT.

SECONDARY OUTCOMES:
Change from baseline in body composition af 2, 6 and 12 weeks | At baseline, 2, 6 and 12 weeks
  As measured by DEXA- and MRI-scanning.
Change from baseline in appetite at 12 weeks | At baseline and 12 weeks
  As measured by food records, controlled diets, meal tests and appetite hormones
Motivational factors for exercise | During and for up to 1½ year after the intervention
  Ethnographic field work
Diameter of t-tubuli in skeletal muscle | At baseline
  As measured in skeletal muscle biopsies by electron and confocal microscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Biomedical Sciences, The University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- See also: Click here for more information about this study: Physical Activity for a Long and Healthy Life — http://fine.ku.dk